CLINICAL TRIAL: NCT05065359
Title: A Randomized, Double-Blinded, Placebo-Controlled, MultipleAscending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Rodatristat Ethyl in Healthy Japanese and Caucasian Subjects
Brief Title: Multiple-Ascending Dose in Japanese Patients Bridging Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altavant Sciences GmbH (Industry)
Collaborators: Altavant Sciences, Inc. (Unknown); Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-1201-1005
Record Dates: First submitted 2021-08-02; First posted 2021-10-04 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: Healthy
Keywords: Pulmonary Arterial Hypertension; PAH
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — rodatristat; BID protein, human

STUDY DESIGN:
Intervention Model Description: Multiple Ascending Dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Rodatristat Ethyl 300 mg BID - Japanese subjects (Experimental)
  Interventions: Drug: Rodatristat Ethyl 300 mg BID
- Placebo match for Rodatristat Ethyl 300 mg BID - Japanese subjects (Placebo Comparator)
  Interventions: Drug: Placebo
- Rodatristat Ethyl 300 mg BID - Caucasian subjects (Experimental)
  Interventions: Drug: Rodatristat Ethyl 300 mg BID
- Placebo match for Rodatristat Ethyl 300 mg BID - Caucasian subjects (Placebo Comparator)
  Interventions: Drug: Placebo
- Rodatristat Ethyl 600 mg BID - Japanese subjects (Experimental)
  Interventions: Drug: Rodatristat Ethyl 600 mg BID
- Placebo match for Rodatristat Ethyl 600 mg BID - Japanese subjects (Placebo Comparator)
  Interventions: Drug: Placebo
- Rodatristat Ethyl 600 mg BID - Caucasian subjects (Experimental)
  Interventions: Drug: Rodatristat Ethyl 600 mg BID
- Placebo match for Rodatristat Ethyl 600 mg BID - Caucasian subjects (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rodatristat Ethyl 300 mg BID — Tablets, oral, 300 mg, BID 14 days
  Arms: Rodatristat Ethyl 300 mg BID - Caucasian subjects; Rodatristat Ethyl 300 mg BID - Japanese subjects
Drug: Rodatristat Ethyl 600 mg BID — Tablets, oral, 600 mg, BID 14 days
  Arms: Rodatristat Ethyl 600 mg BID - Caucasian subjects; Rodatristat Ethyl 600 mg BID - Japanese subjects
Drug: Placebo — Tablets, oral, 0 mg, BID for 14 days
  Arms: Placebo match for Rodatristat Ethyl 300 mg BID - Caucasian subjects; Placebo match for Rodatristat Ethyl 300 mg BID - Japanese subjects; Placebo match for Rodatristat Ethyl 600 mg BID - Caucasian subjects; Placebo match for Rodatristat Ethyl 600 mg BID - Japanese subjects

SUMMARY:
This study is a randomized, placebo-controlled, multiple-ascending dose study in healthy Japanese and Caucasian subjects.

DETAILED DESCRIPTION:
This study is a randomized, placebo-controlled, multiple-ascending dose study in healthy Japanese and Caucasian subjects. Two dose levels of rodatristat ethyl, 300 mg twice daily (BID) and 600 mg BID multiple doses (with a single dose lead in), will be explored in an ascending dose fashion with a safety review in between (Figure 1 below). Approximately 48 subjects will be enrolled in 4 cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females aged 18 to 55 years, inclusive
* A male subject is eligible to participate if he does not have a female partner who is pregnant or who intends to become pregnant during the study. Male subjects must agree to use contraception starting at Screening, during the treatment period, and for at least 100 days after the last dose of Investigational Product (IP), and refrain from donating sperm during this period.
* Female subjects of childbearing potential must agree to use contraception starting at Screening, during the treatment period, and for at least 30 days after the last dose of IP.
* Body mass index (BMI) ≥ 18 kg/m2 and ≤ 32 kg/m2 at Screening
* Japanese subjects must have been born in Japan and not have lived outside of Japan > 10 years at the time of Screening, have both parents and grandparents of ethnic Japanese origin, and have not significantly modified their diets since leaving Japan.
* Caucasian subjects must be of European or Latin American descent (i.e., White).
* Capable of giving signed informed consent, able to understand and comply with protocol requirements, instructions, and protocol related restrictions, and likely to complete the study as planned.

Exclusion Criteria:

* Any known pre-existing medical or psychiatric condition that could interfere with the subject's ability to provide informed consent or participate in study conduct, or that may confound study findings including, but not limited to a history of clinically significant gastrointestinal, hematologic, renal, hepatic, bronchopulmonary, neurological, psychiatric, or cardiovascular disease
* a. History of Gilbert's Syndrome
* b. History of depression
* c. History of any allergy that, in the opinion of the Investigator, contraindicates participation in the trial
* Any positive finding on the Columbia-Suicide Severity Rating Scale (C-SSRS).
* Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at Screening) of 50 mL to 499 mL of blood within 30 days or more than 499 mL within 56 days prior to Day 1
* Participation in an investigational drug, vaccine, or device study within 30 days before IP administration or 90 days for a biologic study
* Evidence of previous myocardial infarction
* a. Any conduction abnormality (including but not specific to atrioventricular block [2nd degree or higher], Wolff Parkinson White syndrome [unless curative ablation treatment]).
* b. Sinus pauses > 3 seconds.
* c. Any significant arrhythmia which, in the opinion of the Investigator and Medical Monitor, will interfere with the safety for the individual subject.
* d. Non-sustained or sustained ventricular tachycardia (≥ 3 consecutive ventricular ectopic beats).
* Abnormal blood pressure, either low (defined as < 90 mmHg systolic and/or < 50 mmHg diastolic) or high (defined as > 140 mmHg systolic and/or > 90 mmHg diastolic)
* Clinically significant abnormalities in laboratory test results (including hepatic and renal panels, complete blood count, coagulation, chemistry panel, and urinalysis)
* a. Positive serology for hepatitis B, hepatitis C virus, or human immunodeficiency virus
* b. Estimated glomerular filtration rate < 80 mL/min/1.73 m2
* c. Aspartate aminotransferase, alanine aminotransferase values greater than 1.5 x upper limit of normal.
* d. Positive urine test for drugs of abuse
* e. Positive alcohol test (breath, saliva, or urine)
* Use of prescription or nonprescription drugs including high dose vitamins, dietary supplements (including St. John's Wort) within 7 days or 5 half-lives of the prescription or nonprescription drug (whichever was longer) prior to the first dose of IP product, unless in the opinion of the Investigator and Sponsor, the medication would not interfere with the study outcomes or compromise subject safety.
* Subject unable to abstain from consumption of tryptophan-rich foods 48 hours prior to admission to the clinic through the Follow-up visit
* Consumption of grapefruit or Seville oranges or their juices within the 7 days prior to dosing until collection of the final PK sample.
* Use of medications associated with QT prolongation within 30 days prior to dosing and during the study. A list of prohibited medications is provided in an appendix to the protocol.
* Subjects unable to abstain from alcohol for 72 hours prior to the start of dosing through collection of their final PK sample
* Subjects with a clinical history of or current alcohol abuse defined as an average weekly intake of more than 21 units for males or 15 units for females (1 unit = 340 mL beer, 115 mL wine, or 43 mL spirits).
* Subjects with a clinical history of or current illicit drug use which, in the opinion of the Investigator, would interfere with the subject's ability to complete the study and could compromise subject safety and/or the results of the study.
* Subjects unable to abstain from caffeine, xanthine, or strenuous exercise for 72 hours prior to dosing until collection of their final PK sample.
* Subjects who have smoked or used tobacco or nicotine-containing products or cannabidiol and related products (in all forms) within 3 months prior to the Screening visit and who are unwilling to refrain from cannabidiol and related products, smoking, tobacco use, or use of nicotine products and all for the entire duration of the study (through the Follow-up visit)
* History of hypersensitivity to rodatristat ethyl, any its components, or any components in the placebo preparation.
* Employed as site personnel directly involved with this study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Safety of rodatristat ethyl by incidence of adverse events | 21 days
  Assessments of adverse events

SECONDARY OUTCOMES:
Single dose AUC(0-∞) | 21 days
  Single dose area under the concentration time curve from time zero (predose-) extrapolated to infinity (AUC(0-∞)) of rodatristat ethyl and metabolite(s).
Single dose AUC(0-t) | 21 days
  Single dose area under the concentration time curve from time zero to the last detectable time point (AUC(0-t)) of rodatristat ethyl and metabolite(s).
Single dose Cmax | 21 days
  Single dose maximum observed concentration (Cmax) of rodatristat ethyl and metabolite(s).
Single dose tmax | 21 days
  Single dose time to maximum concentration (tmax) of rodatristat ethyl and metabolite(s).
Single dose t½ | 21 days
  Single dose elimination half-life (t½) of rodatristat ethyl and metabolite(s).
Steady state tmax | 21 days
  Steady-state tmax of rodatristat ethyl and metabolite(s).
Steady state Cmax | 21 days
  Steady-state Cmax of rodatristat ethyl and metabolite(s).
Steady state Cτ | 21 days
  Steady-state concentration at end of dosing interval (Cτ) of rodatristat ethyl and metabolite(s).
Steady state Cavg | 21 days
  Steady-state average concentration at steady state (Cavg) of rodatristat ethyl and metabolite(s).
Steady state AUC(0-τ) | 21 days
  Steady-state area under the concentration-time curve over the dosing interval at steady-state (AUC(0-τ)) of rodatristat ethyl and metabolite(s).
Steady state t½ | 21 days
  Steady-state t½ of rodatristat ethyl and metabolite(s).
Pharmacodynamic assessment - change from baseline in 5-HIAA concentrations | 21 days
  PD as assessed by the change from baseline in 5-hydroxyindoleacedtic acid (5-HIAA) concentrations (plasma and 24-hour urinary excretion)

CONTACTS AND LOCATIONS:
Locations (1):
- California Clinical Trials Medical Group (CCTMG), Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No